CLINICAL TRIAL: NCT02452918
Title: An Open-Label Study to Evaluate the Safety of a Single 1200 mg IV Dose of Orbactiv (Oritavancin) in Subjects on Concomitant Chronic Warfarin Therapy Being Treated For Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Brief Title: A Study to Evaluate the Safety of a Single Intravenous (IV) Dose of Orbactiv (Oritavancin) in Participants on Chronic Warfarin Therapy Being Treated For Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-ORI-14-03
Record Dates: First submitted 2015-05-13; First posted 2015-05-25 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Acute Bacterial Skin and Skin Structure Infection
Keywords: skin infection
MeSH Terms: conditions — Cellulitis | interventions — oritavancin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oritavancin 1200 mg Without Concomitant Warfarin Therapy (Experimental): Oritavancin as a single 1200 mg IV dose administered over 3 hours in participants with ABSSSI who were not on concomitant warfarin therapy
  Interventions: Drug: Oritavancin
- Oritavancin 1200 mg With Concomitant Warfarin Therapy (Experimental): Oritavancin as a single 1200 mg IV dose administered over 3 hours in participants with ABSSSI who were on concomitant warfarin therapy at a standard dose and dosing schedule
  Interventions: Drug: Oritavancin; Drug: Warfarin

INTERVENTIONS:
Drug: Oritavancin — Administered intravenously
  Other Names: Orbactiv
Drug: Warfarin — Administered as a concomitant medication at a standard dose and dosing schedule
  Arms: Oritavancin 1200 mg With Concomitant Warfarin Therapy

SUMMARY:
This was a Phase 4, multicenter, open-label safety study of a single 1200 milligrams (mg) IV infusion of oritavancin in adult participants on chronic warfarin with acute bacterial skin and skin structure infection (ABSSSI) suspected or proven to be caused by Gram-positive pathogens.

An additional group of participants with ABSSSI, who were not on concomitant warfarin therapy, were also enrolled to obtain additional information following a single dose of oritavancin administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ABSSSI (wound infection, cellulitis/erysipelas, or cutaneous abscess) suspected or confirmed to be caused by a Gram-positive pathogen requiring IV therapy
* Must be currently being treated with chronic warfarin therapy* *Participants in the non-warfarin group are not required to be on chronic warfarin therapy.

Exclusion Criteria:

* Known or suspected bacteremia, sepsis or refractory shock
* Participants who are likely to need treatment with IV heparin within 48 hours
* Significant or life-threatening condition
* Women who are pregnant or nursing
* Receiving chronic systemic immunosuppressive therapy such as chemotherapy or prednisone
* CD4 count <200 cells/mm^3 in participants with known human immunodeficiency virus or acquired immune deficiency syndrome
* Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- Somers Point, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oritavancin 1200 mg Without Concomitant Warfarin Therapy: Oritavancin as a single 1200 mg intravenous (IV) dose administered over 3 hours in participants with acute bacterial skin and skin structure infection (ABSSSI) who were not on concomitant warfarin therapy
- Oritavancin 1200 mg With Concomitant Warfarin Therapy: Oritavancin as a single 1200 mg IV dose administered over 3 hours in participants with ABSSSI who were on concomitant warfarin therapy
Period: Overall Study
Arm/Group | Oritavancin 1200 mg Without Concomitant Warfarin Therapy | Oritavancin 1200 mg With Concomitant Warfarin Therapy
Started | 15 | 2
Received at Least 1 Dose of Study Drug | 15 | 2
Completed | 15 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all participants who were screened and enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Oritavancin 1200 mg Without Concomitant Warfarin Therapy | Oritavancin 1200 mg With Concomitant Warfarin Therapy | Total
Number analyzed (Participants) | 15 | 2 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 0 | 14
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 2 | 16
  Black or African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment, including abnormal vital signs or laboratory assessments. An SAE was defined as any untoward medical occurrence that at any dose resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 2 weeks after first administration of oritavancin
Population: Safety analysis population included all participants who were dosed with IV oritavancin
Measure: Count of Participants; unit: Participants
Arm/Group | Oritavancin 1200 mg Without Concomitant Warfarin Therapy | Oritavancin 1200 mg With Concomitant Warfarin Therapy
Number analyzed (Participants) | 15 | 2
Participants
  At least 1 AE | 2 | 1
  At least 1 SAE | 0 | 0

2. Secondary Outcome: Number of Participants With a Clinical Response of Cure
Description: Participants were classified by investigator assessment as "success" for clinical response of cure if all of the following were met: cessation of spread or reduction of the lesion; resolution (absence) of fever (temperature less than 37.7° Celsius); no rescue antibiotic medication; complete or nearly complete resolution of baseline signs and symptoms of the primary infection such that no further treatment with antibiotics was needed.
Time Frame: At 48 to 72 hours after start of oritavancin dose and at Day 7
Population: Safety analysis population included all participants who were dosed with IV oritavancin
Measure: Count of Participants; unit: Participants
Arm/Group | Oritavancin 1200 mg Without Concomitant Warfarin Therapy | Oritavancin 1200 mg With Concomitant Warfarin Therapy
Number analyzed (Participants) | 15 | 2
Participants | 15 | 2

ADVERSE EVENTS:
Time Frame: Up to 2 weeks after first administration of oritavancin
Description: Safety analysis population included all participants who were dosed with IV oritavancin.
Arm/Group | Oritavancin 1200 mg Without Concomitant Warfarin Therapy | Oritavancin 1200 mg With Concomitant Warfarin Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/2
Other Adverse Events (participants affected / at risk) | 2/15 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oritavancin 1200 mg Without Concomitant Warfarin Therapy (N=15) | Oritavancin 1200 mg With Concomitant Warfarin Therapy (N=2)
Infusion site phlebitis (General disorders) | 1 | 0
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02452918/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT02452918/SAP_001.pdf